CLINICAL TRIAL: NCT05733533
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Study of Efficacy and Safety of HRS-2261 in Refractory Chronic Cough
Brief Title: A Study to Assess the Efficacy and Tolerance of HRS-2261 in Subjects With Refractory Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2261-201
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-2261 oral tablet (Experimental)
  Interventions: Drug: HRS-2261 oral tablet
- Matching placebo to HRS-2261 (Placebo Comparator)
  Interventions: Drug: Matching placebo to HRS-2261

INTERVENTIONS:
Drug: HRS-2261 oral tablet — HRS-2261 oral tablet, oral, BID
  Arms: HRS-2261 oral tablet
Drug: Matching placebo to HRS-2261 — Matching placebo to HRS-2261, oral, BID
  Arms: Matching placebo to HRS-2261

SUMMARY:
This is a phase II study that will investigate the efficacy, safety and tolerability of HRS-2261 in subjects with refractory chronic cough using a double blind, placebo controlled, randomized study design.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. Diagnosed with refractory chronic cough or chronic cough of unknown cause, with a course of disease lasting more than 1 year;
3. Within 5 years prior to screening and after the onset of chronic cough, chest imaging did not reveal any significant abnormalities that the investigators considered to cause chronic cough or any other clinically significant lung disease;
4. VAS scores of cough severity in screening period and baseline period ≥ 40 mm;
5. Subjects receiving medication for pre-existing underlying conditions prior to the screening period should stabilize the corresponding dose for at least 8 weeks prior to screening;
6. Take effective contraceptive measures;
7. Voluntarily sign informed consent to participate in this study;
8. Willing and able to comply with all protocol requirements, including demonstrating the ability to comply with study procedures prior to random assignment.

Exclusion Criteria:

1. Patients diagnosed with chronic obstructive pulmonary disease (COPD), bronchiectasis, idiopathic pulmonary fibrosis (IPF), and endobronchial tuberculosis;
2. Patients with a history of chronic bronchitis;
3. Patients with a history of upper or lower respiratory tract infection, or acute exacerbation of respiratory disease, or significant changes in chest imaging within 4 weeks prior to baseline period;
4. Current smokers, smokers who have quit smoking (within 6 months), or former smokers who consume more than 20 packs of cigarettes per year;
5. Those with abnormal taste within 3 months prior to previous diagnosis or screening;
6. Malignant disease within 5 years or less before signing the informed consent, except for basal cell or squamous cell skin cancer or cervical cancer in situ after appropriate treatment;
7. Currently taking or having taken an angiotensin-converting enzyme inhibitor in the 3 months prior to screening;
8. Those who are currently taking or have used any antitussive medication within the week prior to screening;
9. Patients who had used oral steroids or antiallergy drugs within 1 week prior to screening;
10. Screening or baseline 1 second rate < 60%;
11. Poorly controlled hypertension;
12. Alanine aminotransferase or aspartate aminotransferase more than 2 times the upper limit of normal in screening period or baseline period;
13. Estimated glomerular filtration rate (eGFR) < 30mL/min/1.73m2 or eGFR≥30mL/min/1.73m2 and <50mL/min/1.73m2 with unstable renal function during screening;
14. Use of systemic immunosuppressants or immunomodulators, or biologics or Th2 cytokine inhibitors within 12 weeks prior to randomization or within 5 half-lives of the drug;
15. A recent history of drug or alcohol abuse or dependence (within the past 1 year);
16. Participants enrolled in clinical trials of any drug or medical device within 3 months prior to screening, or within 5 half-lives of test drugs before screening, whichever is longer;
17. Any past or present circumstances, determined by the investigator or sponsor, make the subject unfit for admission to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in visual analog Scale (VAS) scores of cough severity after 4 weeks of treatment (Day 28) | Baseline (Day-1)，Day 28

SECONDARY OUTCOMES:
Changes from baseline in patients' overall Impression of Change (PGIC) scale scores after week 1, 2, 3 and 4 of treatment (Day 7, Day 14, Day 21, Day 28) | Day 7, Day 14, Day 21, Day 28
Changes from baseline in the total score of the Leicester Cough Questionnaire (LCQ), which assessed cough-specific quality of life, at 2 and 4 weeks after treatment (Day 14, Day 28) | Baseline (Day-1), Day 14, Day 28
Changes from baseline in the simple cough severity score (CET) at week 1, 2, 3, and 4 after treatment (Day 7, Day 14, Day 21, Day 28) | Day 7, Day 14, Day 21, Day 28
Incidence and severity of any adverse events (AE) | up to 6 weeks (Day 42)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided